CLINICAL TRIAL: NCT06714877
Title: A Single-center, Prospective, Randomized Controlled Trial Evaluating Type a Botulinum Toxin Injection and Prism Therapy for the Treatment of Acute Acquired Concomitant Esotropia
Brief Title: Botulinum Toxin Injection Versus Prism Treatment in Small-angle Acute Acquired Concomitant Esotropia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-BTXAACE
Record Dates: First submitted 2024-12-02; First posted 2024-12-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Esotropia
Keywords: Acute Acquired Concomitant Esotropia; Treatment; Botulinum Toxin Injection
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prism treatment group (Active Comparator): prism treatment
  Interventions: Other: prism treatment group
- botulinum toxin group (Experimental): botulinum toxin injection
  Interventions: Procedure: botulinum toxin group

INTERVENTIONS:
Other: prism treatment group — wearing prism glasses
  Arms: prism treatment group
Procedure: botulinum toxin group — botulinum toxin injection
  Arms: botulinum toxin group

SUMMARY:
This is a single-center, prospective, randomized controlled trial evaluating type A botulinum toxin injection and prism therapy for the treatment of small-angle acute acquired concomitant esotropia.

Specific Aim 1 (Primary): To compare the reduction of deviation angle and improvement of diplopia symptoms between botulinum toxin injection and prism therapy for the treatment of small-angle acute acquired concomitant esotropia.

Specific Aim 2 (Secondary): To compare the improvement of visual functions between botulinum toxin injection and prism therapy for the treatment of small-angle acute acquired concomitant esotropia.

DETAILED DESCRIPTION:
Acute acquired concomitant esotropia (AACE) belongs to the category of concomitant strabismus, which manifests as sudden onset, often accompanied by diplopia, and no change in the strabismus angle of each eye position. In recent years, with the increase in the use of smartphones and other screen devices, the incidence of AACE has been on the rise. Commonly used treatments in clinical practice include surgical treatment, botulinum toxin injection, and prism treatment. Patients with large deviation angel generally require surgical intervention to fundamentally correct their eye position and eliminate diplopia, but surgical treatment requires waiting for six months and can only be performed after the patient's strabismus degree is stable, and there is a risk of intraoperative trauma and secondary surgery. Patients with early and small-angle strabismus often choose prism treatment.

The principle of prism treatment is light refraction. After the light is refracted through the prism, it falls on the fovea of the strabismic eye, eliminating diplopia. In the treatment of AACE, the main target population of prisms is patients with mild strabismus (the strabismus angle is usually less than 25 PD. Wearing prisms can eliminate diplopia and relieve related symptoms, but it does not really correct the patient's strabismus problem.

Botulinum toxin treatment is to inject botulinum toxin type A into the medial rectus muscle to weaken the muscle strength and improve strabismus. Although it has not been widely used in clinical practice, a large number of studies have compared the efficacy of botulinum toxin treatment and surgical treatment. Some studies have found that the efficacy of the two is equivalent, which indicates that botulinum toxin treatment may be a good treatment option for AACE. Botulinum toxin treatment has the advantages of simple operation, low patient cooperation requirements, fast recovery, low trauma, and low treatment cost. It may become a treatment option for patients with small angle AACE. There are also reports that temporary ptosis and overcorrection may occur after botulinum toxin injection. The safety of botulinum toxin injection treatment also needs to be explored. However, existing studies have not fully explored the effectiveness and safety of botulinum toxin in the treatment of small-angle AACE, nor have studies compared the therapeutic effects of prisms and botulinum toxin on small-angle AACE.

In order to better guide clinical practice, we conducted this prospective cohort study to objectively evaluate and compare the therapeutic effects of botulinum toxin and prism treatment on AACE. It is expected that the results of the study will provide more treatment options for AACE patients and provide important guidance for the clinical selection of appropriate methods to treat small-angle AACE.

ELIGIBILITY:
Inclusion Criteria:

1. acute acquired concomitant esotropia diagnosis (sudden onset of esotropia or diplopia, no significant change in the degree of strabismus in each eye position, and no limitation in eye movement)
2. strabismus angle ≤ 25PD
3. best corrected visual acuity of both eyes ≥ 1.0
4. intracranial disease is excluded by cranial CT or magnetic resonance imaging

Exclusion Criteria:

1. reduction of strabismus angle by more than 10 prism diopters after refractive correction
2. history of other ocular diseases or ocular surgeries
3. presence of organic brain lesions or systemic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
strabismus angle | Before treatment, 1 week, 1 month, 3 months, 6 months after treatment
  using prism cover test to evaluate the reduction of strabismus angle

SECONDARY OUTCOMES:
stereopsis | Before treatment, 1 week, 1 month, 3 months, 6 months after treatment
  using randot stereotest to evaluate the improvement of stereopsis

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wen, MD, PhD, Study Chair — Eye & ENT Hospital of Fudan University, Shanghai, China
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it's better to protect the publication potential.